CLINICAL TRIAL: NCT01437475
Title: Efficiency of the Novel Hepatitis B Vaccine Sci-B-Vac in HIV Positive Patients, a Prospective Cohort Study
Brief Title: Efficiency of the Hepatitis B Sci-B-Vac Vaccine in HIV Positive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: SciGen, Israel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-11-DA-0277-CITL
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: HIV
Keywords: HBV; HIV; Immunization; HBV Immunization rate among HIV positive individuals
MeSH Terms: interventions — Pre-S vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sci-B-Vac (Experimental): The study involves only one, open label arm. Rate of immunization will be compared to results obtained using the ENGERIX B vaccine among HIV positive persons in formerly published, historical cohorts.
  Interventions: Biological: Sci-B-Vac

INTERVENTIONS:
Biological: Sci-B-Vac — 10 microgram/ml hepatitis B surface antigen, 1 ml given intramuscularly

SUMMARY:
HBV vaccination is of paramount importance among HIV positive persons due to an increased risk of infection and disease progression. The most widely used ENGERIX B vaccine reaches a lower rate of vaccination (20-70%) among HIV positive vaccinees (compared to over 90% in the normal population). Sci-B-Vac is novel vaccine containing 3 antigens and is therefore more immunogenic (as opposed to one in ENGERIX B). Its use has been associated with higher and more rapid vaccination rates. Therefore, it has a theoretical advantage in HIV positive individuals.

DETAILED DESCRIPTION:
A cohort of 100 HIV positive, HBV negative individuals who have not been vaccinated against HBV before will be prospectively given 3 doses of Sci-B-Vac at 0, 1 and 6 months. HBV antibodies will be checked one month after every dose given.

ELIGIBILITY:
Inclusion Criteria:

* HBV negative
* HIV positive individuals
* Above the age of 18
* Treated at the TASMC Aids clinic, who have signed and informed consent and have never been vaccinated against HBV before

Exclusion Criteria:

* Pregnant women
* HBV positivity
* Previous HBV vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-03 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
HBV immunization rate after 1, 2 and 3rd dose of Sci-B-Vac | 12 months
  HBV Surface antibodies will be obtained one month after each Sci-B-Vac dose for each vaccinee. Rate and rapidity of immunization will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Turner, MD, Study Chair — Tel-Aviv Sourasky Medical Center; Danny Alon, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Dan Turner, Tel Aviv, Israel

REFERENCES:
- [Background] 1. R. van den Berg, I. van Hoogstraten and M. van Agtmael. Non-Responsiveness to Hepatitis B Vaccination in HIV Seropositive Patients; Possible causes and solutions. AIDS Rev. 2009;11:157-65. 2. O. Launay, D. van der Vilet, A. Rosenberg et al. Safety and Immunogenicity of 4 Intramuscular double doses and 4 intradermal low doses vs standard hepatitis B vaccine regimen in adults with HIV-1. JAMA, 2001; Vol 35. No.14:1432-1440. 3. Petit NN, DePestel DD, Malani PN et al. Factors associated with seroconversion after standard dose hepatitis B vaccination and high dose revaccination among HIV-infected patients. HIV Clin Trials. 2010 Nov-Dec;11(6):332-9. 4. MY Shapira, E. Zeira, R. Rapid seroprotection against hepatitis B following the first dose of a Pre-S1/Pre-S2/S vaccine. Journal of Hepatology 34 (2001); 123-127. 5. SM Fiedler, U. Dahmen, H. Grosse-Wilde et al. Cellular and humoral immune response to a third generation hepatitis B vaccine. Journal of viral hepatitis. 2007, 14: 592-598. 6. Paitoonpong L., Suankratay C. Immunological response to hepatitis B vaccination in patients with Aids and virological response to HAART. Scan J Infect Dis. 2008;40(1):54-8. 7. Laurence J. Hepatitis A and B immunizations of individuals infected with HIV. Am J Med. 2005;118 (Suppl. 10A: 75-93s). 8. Pasnicha N, Datta U, Chawla Y et al. Immune responses in patients with HIV infection after vaccination with recombinant hepatitis B virus vaccine. BMC Infec Dis 2008;8:85.